CLINICAL TRIAL: NCT06607601
Title: CARE Initiative Study: Real-world Emulation of the PALOMA-2 Comparative Effectiveness Trial of Palbociclib and Letrozole vs. Placebo and Letrozole for the First-line Treatment of ER+/HER2- Advanced Breast Cancer
Brief Title: CARE Initiative: Real-world Emulation of the PALOMA-2 Trial
Status: Completed | Type: Observational
Sponsor: Aetion, Inc. (Other)
Collaborators: AbbVie (Industry); Amgen (Industry); AstraZeneca (Industry); Bayer (Industry); Gilead Sciences (Industry); Janssen, LP (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: DS3-PALOMA2
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Breast Cancer
Keywords: real-world evidence; real-world data; oncology; pharmacoepidemiology; comparative effectiveness research; trial emulation
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Exposed: Patients initiating treatment with palbociclib and letrozole as first-line treatment for metastatic ER+/HER2- breast cancer
  Interventions: Drug: Palbociclib; Drug: Letrozole
- Comparator: Patients initiating treatment with letrozole as first-line treatment for metastatic ER+/HER2- breast cancer
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — Treatment information in the electronic health record indicates initiation of palbociclib after metastatic diagnosis
  Groups: Exposed
Drug: Letrozole — Treatment information in the electronic health record indicates initiation of letrozole after metastatic diagnosis

SUMMARY:
The goal of this non-interventional study is to emulate the PALOMA-2 randomized controlled trial of palbociclib as first-line therapy in patients with estrogen receptor-positive (ER+)/human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer using real-world, electronic health record data. The main questions this study aims to answer are:

1. Do patients with metastatic ER+/HER2- breast cancer treated with palbociclib and letrozole have improved real-world progression-free survival (rwPFS) compared with patients treated with letrozole alone?
2. How do the results of this non-interventional study compare to those of the PALOMA-2 randomized controlled trial?

DETAILED DESCRIPTION:
The Coalition to Advance Real-World Evidence through Randomized Controlled Trial Emulation (CARE) Initiative is a program designed to build an empirical evidence base for the use of real-world data (RWD) in clinical and regulatory decision-making. Using randomized controlled trials (RCT) as a benchmark for causal effect estimates, a series of RCT emulations will be conducted across varying trials, real world data sources, and study design elements to better understand under what conditions non-interventional studies, using data generated during routine clinical care, can provide reliable conclusions about drug effectiveness.

In this study, real-world electronic health record (EHR) data will be used to emulate the Palbociclib: Ongoing Trials in the Management of Breast Cancer (PALOMA-2) efficacy trial of palbociclib as first-line therapy in patients with estrogen receptor-positive (ER+)/human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer.2 Similarly to the PALOMA-2 trial, this study will compare real-world progression-free survival (rwPFS) between patients who initiate palbociclib and letrozole and those initiating letrozole alone.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis
* Histology not indicative of non-adenocarcinoma histologies
* Metastatic disease
* Estrogen-receptor positive (ER+)
* No prior systemic treatment for metastatic breast cancer
* Post-menopausal
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2 or missing or Karnofsky performance status >=50 or missing
* No lab results indicating inadequate organ function, as defined in the PALOMA-2 RCT protocol

Exclusion Criteria:

* Human epidermal growth factor receptor 2 (HER2) positive tumor
* Diagnosis of brain, central nervous system, and/or spinal cord metastases
* Neoadjuvant or adjuvant treatment with anastrozole or letrozole ≤12 months before metastatic diagnosis
* Prior treatment with treatment with ribociclib, abemaciclib, or palbociclib
* Treatment with a CYP3A4 inhibitor or inducer or drugs known to prolong the QT interval, as specified in the PALOMA-2 trial protocol, in the 7 days prior to study treatment initiation
* Anti-cancer therapy or major cancer-related surgery within 2 weeks before study treatment initiation
* Diagnosis of a second primary malignancy within 3 years prior to study treatment initiation
* Diagnosis of long or short QT syndrome, Brugada syndrome, QTc prolongation, or Torsade de Pointes
* Diagnosis of hypocalcemia, hypokalemia, or hypomagnesemia
* Diagnosis of myocardial infarction, angina, ongoing cardiac dysrhythmias, atrial fibrillation, congestive heart failure, cerebral infarction, transient ischemic attack, or pulmonary embolism in the 6 months prior to study treatment initiation
* Diagnosis of inflammatory bowel disease chronic diarrhea, or short bowel syndrome
* Diagnosis of human immunodeficiency virus infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified in the electronic health record data source with metastatic ER+/HER2- breast cancer initiating treatment with the study drugs (palbociclib, letrozole)
Sampling Method: Non-Probability Sample
Enrollment: 724 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Real-world progression-free survival (rwPFS) | From study treatment initiation until the date of disease progression, death from any cause or censoring, whichever came first, assessed up to 33 months.
  Time from study treatment initiation to disease progression or death

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT06607601/Prot_SAP_000.pdf